CLINICAL TRIAL: NCT03806933
Title: A Prospective, Randomized, Double-blind, Multicenter Study to Investigate the Safety and Duration of Effect of Different NT 201 Dose Groups Following the Treatment of Glabellar Frown Lines
Brief Title: Study to Investigate the Safety and Duration of Effect of Different Botulinum Toxin A (NT 201) Dose Groups Following the Treatment of Glabellar Frown Lines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merz Aesthetics GmbH (Industry)
Collaborators: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M602011015; 2018-002743-28 (EudraCT Number)
Record Dates: First submitted 2019-01-15; First posted 2019-01-16 (Actual); Results first posted 2023-10-04 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Moderate to Severe Glabellar Frown Lines
MeSH Terms: interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- NT 201 Dose group 1 (Experimental): Stage 1 and 2. Intramuscular injection into the glabellar area.
  Interventions: Drug: NT 201
- NT 201 Dose group 2 (Experimental): Stage 1. Intramuscular injection into the glabellar area.
  Interventions: Drug: NT 201
- NT 201 Dose group 3 (Experimental): Stage 1. Intramuscular injection into the glabellar area.
  Interventions: Drug: NT 201
- NT 201 Dose group 4 (Experimental): Stage 2. Intramuscular injection into the glabellar area.
  Interventions: Drug: NT 201
- NT 201 Dose group 5 (Experimental): Open Label Extension Period. Intramuscular injection into the glabellar area.
  Interventions: Drug: NT 201

INTERVENTIONS:
Drug: NT 201 — Clostridium Botulinum neurotoxin Type A free from complexing proteins. Solution for injection prepared by reconstitution of powder with 0.9% unpreserved Sodium Chloride (NaCl).
  Other Names: IncobotulinumtoxinA; Xeomin; Botulinum toxin type A (150 kiloDalton), free from complexing proteins

SUMMARY:
The purpose of the study is to investigate the safety and duration of effect following different doses of Botulinum Toxin A (NT 201) in the treatment of glabellar frown lines (GFL).

DETAILED DESCRIPTION:
This prospective, randomized, double-blind, multi-Center clinical study consists of a two stage experimental main period comparing different dose groups, followed by an optional open-label extension period (20 Units follow-up treatment).

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant 18 years or over.
* Moderate (score=2) to severe (score=3) GFL at maximum frown as assessed by investigator on the 4-point facial wrinkle scale (FWS).
* Moderate (score=2) to severe (score=3) GFL at maximum frown as assessed by participant on the 4-point FWS.

Exclusion Criteria:

* Previous treatment with Botulinum neurotoxin (BoNT) of any serotype in the facial area within the last 12 months before injection.
* Previous treatment with any facial cosmetic procedure (example, chemical peeling, photo rejuvenation, mesotherapy, photodynamic therapy, laser treatment, tattooing of eyebrows) in the glabellar area within the last 12 months before injection.
* Previous treatment with any biodegradable filler in the glabellar area within the last 12 months before injection.
* Inability to substantially reduce GFL by physically spreading them apart as assessed by the investigator.
* Excessively thick sebaceous skin or hypertrophic muscles in the upper third part of the face.
* Any surgery or scars in the glabellar area.
* Marked facial asymmetry.
* Eyelid ptosis.
* Marked brow ptosis and/or dermatochalasis.
* Ongoing severe or unstable medical conditions, example, systemic infection, or pulmonary disease, at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz Pharmaceuticals GmbH
Locations (9):
- United States (5):
  - Clinical Testing of Beverly Hills, Merz Investigational Site #0010395, Encino, California
  - Medical Associates Inc., Merz Investigational Site #0010435, Newport Beach, California
  - Cosmetic Laser Dermatology, Merz Investigational Site #0010321, San Diego, California
  - The Maas Clinics, Merz Investigational Site #0010338, San Francisco, California
  - Tennessee Clinical Research Center, Merz Investigational Site #0010097, Nashville, Tennessee
- Germany (4):
  - Privatpraxis für Dermatologie und Ästhetische Medizin, Merz Investigational Site #0490306, Berlin
  - Universität Hamburg, Fachrichtung Kosmetik und Körperpflege, Merz Investigational Site #0490095, Hamburg
  - Dermatologische Gemeinschaftspraxis Dr. Prager und Partner, Merz Investigational Site #0490345, Hamburg
  - Skin & Laser Center, Merz Investigational Site #0490362, Potsdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kerscher M, Fabi S, Fischer T, Gold M, Joseph J, Prager W, Rzany B, Yoelin S, Roll S, Klein G, Maas C. IncobotulinumtoxinA Demonstrates Safety and Prolonged Duration of Effect in a Dose-Ranging Study for Glabellar Lines. J Drugs Dermatol. 2021 Oct 1;20(10):1052-1060. doi: 10.36849/JDD.6377. PMID 34636520

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 9 sites in Germany and the United States from 23 January 2019 to 8 October 2020. Out of 256 participants, 15 participants were screen failures and 241 participants were enrolled and randomized in the study. Study had 2 periods: Main Period (MP) and an optional Open-label Extension (OLEX) Period. As planned, combined safety data for MP and OLEX Period was reported.
Pre-assignment Details: In MP, Stage 1, participants received NT 201: 20 unit (U), 50 U or 75 U. Based on safety data of Stage 1, Stage 2 was started, and participants received NT 201 20 U or 100 U. After completion of MP, participants had the opportunity to receive an optional follow-up treatment with NT 201 20 U in OLEX period. As planned, 20 U group data from Stages 1 and 2 were pooled.
Groups:
- Stage 1 and 2 Pooled: NT 201 20 U: Participants from Stages 1 and 2 received NT 201 20 U, powder for solution for injection, intramuscularly with the total amount of 0.25 milliliter (mL) injected into the glabellar area in equal aliquots administered to 5 injection sites (0.05 mL per injection site) on Day 1 of MP. This arm consisted of pooled data of all participants who received NT 201 20 U in Stages 1 and 2 of MP. Participants had the opportunity to receive an optional follow-up treatment with the dose of NT 201 20 U with the total amount of 0.5 mL injected into the glabellar area in equal aliquots administered to 5 injection sites (0.1 mL per injection site) in the OLEX period.
- NT 201 50 U: Participants from Stage 1 received NT 201 50 U, powder for solution for injection, intramuscularly with the total amount of 0.25 mL injected into the glabellar area in equal aliquots administered to 5 injection sites (0.05 mL per injection site) on Day 1 of MP. Participants had the opportunity to receive an optional follow-up treatment with the dose of NT 201 20 U with the total amount of 0.5 mL injected into the glabellar area in equal aliquots administered to 5 injection sites (0.1 mL per injection site) in the OLEX period.
- NT 201 75 U: Participants from Stage 1 received NT 201 75 U, powder for solution for injection, intramuscularly with the total amount of 0.25 mL injected into the glabellar area in equal aliquots administered to 5 injection sites (0.05 mL per injection site) on Day 1 of MP. Participants had the opportunity to receive an optional follow-up treatment with the dose of NT 201 20 U with the total amount of 0.5 mL injected into the glabellar area in equal aliquots administered to 5 injection sites (0.1 mL per injection site) in the OLEX period.
- NT 201 100 U: Participants from Stage 2 received NT 201 100 U, powder for solution for injection, intramuscularly with the total amount of 0.25 mL injected into the glabellar area in equal aliquots administered to 5 injection sites (0.05 mL per injection site) on Day 1 of MP. Participants had the opportunity to receive an optional follow-up treatment with the dose of NT 201 20 U with the total amount of 0.5 mL injected into the glabellar area in equal aliquots administered to 5 injection sites (0.1 mL per injection site) in the OLEX period.
Period: Main Period
Arm/Group | Stage 1 and 2 Pooled: NT 201 20 U | NT 201 50 U | NT 201 75 U | NT 201 100 U
Started | 61 | 60 | 61 | 59
Safety Evaluation Set (SES) (One participant randomized to NT 201 100 U dose group was actually treated with NT 201 20 U. The participant was re-assigned to the Pooled: NT 201 20 U dose group for safety analyses.) | 62 | 60 | 61 | 58
Completed | 57 | 57 | 59 | 56
Not Completed | 4 | 3 | 2 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 2
Not completed — Lost to Follow-up | 2 | 2 | 0 | 0
Period: OLEX Period
Arm/Group | Stage 1 and 2 Pooled: NT 201 20 U | NT 201 50 U | NT 201 75 U | NT 201 100 U
Started | 52 (Only participants who relapsed to baseline status of their glabellar frown lines (GFL) in the MP and completed the MP had the opportunity to receive optional follow-up treatment; those receiving optional treatment were entered in the OLEX period.) | 53 (Only participants who relapsed to baseline status of their glabellar frown lines (GFL) in the MP and completed the MP had the opportunity to receive optional follow-up treatment; those receiving optional treatment were entered in the OLEX period.) | 56 (Only participants who relapsed to baseline status of their glabellar frown lines (GFL) in the MP and completed the MP had the opportunity to receive optional follow-up treatment; those receiving optional treatment were entered in the OLEX period.) | 50 (Only participants who relapsed to baseline status of their glabellar frown lines (GFL) in the MP and completed the MP had the opportunity to receive optional follow-up treatment; those receiving optional treatment were entered in the OLEX period.)
Completed | 52 | 53 | 56 | 49
Not Completed | 0 | 0 | 0 | 1
Not completed — Due to coronavirus disease (COVID) 19 pandemic | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) was subset of participants exposed to study medication for whom any efficacy variable was available.
Groups:
- Stage 1 and 2 Pooled: NT 201 20 U: Participants from Stages 1 and 2 received NT 201 20 U, powder for solution for injection, intramuscularly with the total amount of 0.25 mL injected into the glabellar area in equal aliquots administered to 5 injection sites (0.05 mL per injection site) on Day 1 of MP. This arm consisted of pooled data of all participants who received NT 201 20 U in Stages 1 and 2 of MP. Participants had the opportunity to receive an optional follow-up treatment with the dose of NT 201 20 U with the total amount of 0.5 mL injected into the glabellar area in equal aliquots administered to 5 injection sites (0.1 mL per injection site) in the OLEX period.
- Total: Total of all reporting groups
Arm/Group | Stage 1 and 2 Pooled: NT 201 20 U | NT 201 50 U | NT 201 75 U | NT 201 100 U | Total
Number analyzed (Participants) | 61 | 60 | 61 | 59 | 241
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (11.43) | 46.9 (10.27) | 49.2 (13.75) | 49.4 (11.19) | 49.4 (11.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 51 | 54 | 50 | 208
  Male | 8 | 9 | 7 | 9 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 9 | 3 | 13 | 28
  Not Hispanic or Latino | 58 | 51 | 58 | 46 | 213
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Facial Wrinkle Scale (FWS) severity at maximum frown as assessed by the investigator [Count of Participants; unit: Participants] — Investigator's FWS assessed status of GFL according to the 4-point severity grades at maximum frown as: 0 (none), 1 (mild), 2 (moderate), 3 (severe). Descriptors of each severity grade for investigator's FWS assessment at maximum frown were as: 0 (no muscle action at all), 1 (some even slight muscle action possible [that is, visible furrows]), 2 (moderately strong muscle action possible [that is, visible muscle bulges]), 3 (strong muscle action possible which may cause local pallor).
  Participants
    Moderate | 8 | 9 | 9 | 8 | 34
    Severe | 53 | 51 | 52 | 51 | 207

OUTCOME MEASURES:

1. Primary Outcome: Duration of Effect Defined as Time Between Treatment and Relapse to Baseline Status Assessed by the Investigator on the FWS
Description: Duration of effect: time between treatment and first occurrence of relapse to baseline status. If no effect was observed, duration of effect was set to 0. Effect: any improvement (at least 1 point) at maximum frown as assessed by investigator on FWS. Investigator's FWS assessed status of GFL according to 4-point severity grades at maximum frown as: 0 (none), 1 (mild), 2 (moderate), 3 (severe). Descriptors of each severity grade for investigator's FWS assessment at maximum frown were as: 0 (no muscle action at all), 1 (some even slight muscle action possible [that is, visible furrows]), 2 (moderately strong muscle action possible [that is, visible muscle bulges]), 3 (strong muscle action possible which may cause local pallor). Duration of effect was analyzed using Kaplan-meier analysis, and 95 percent (%) confidence interval (CI) were calculated using log-log transformation.
Time Frame: From the time of first treatment up to Day 360
Population: The FAS was subset of participants exposed to study medication for whom any efficacy variable was available.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Stage 1 and 2 Pooled: NT 201 20 U | NT 201 50 U | NT 201 75 U | NT 201 100 U
Number analyzed (Participants) | 61 | 60 | 61 | 59
days | 175 [142 to 185] | 185 [182 to 205] | 210 [182 to 217] | 215 [183 to 237]
Statistical Analysis 1: Comparison: Stage 1 and 2 Pooled: NT 201 20 U vs NT 201 50 U; Test type: Other; p = 0.881, Wald Chi-square test — P-values were based on Wald Chi-Square tests for hazard ratios; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.7 to 1.51] — Hazard ratio (HR) was estimated using a Cox proportional hazards regression model. 95% CIs were calculated based on individual Wald tests
Statistical Analysis 2: Comparison: Stage 1 and 2 Pooled: NT 201 20 U vs NT 201 75 U; Test type: Other; p = 0.089, Wald Chi-square test — P-values were based on Wald Chi-Square tests for hazard ratios; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.49 to 1.05] — HR was estimated using a Cox proportional hazards regression model. 95% CIs were calculated based on individual Wald tests
Statistical Analysis 3: Comparison: Stage 1 and 2 Pooled: NT 201 20 U vs NT 201 100 U; Test type: Other; p = 0.0035, Wald Chi-square test; P-values were based on Wald Chi-Square tests for hazard ratios; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.38 to 0.83] — [estimate comment as in outcome 1, analysis 2]

2. Primary Outcome: Number of Participants With at Least One Treatment-emergent Adverse Event (TEAE)
Time Frame: From the time of first treatment up to Day 390
Population: The SES was the subset of all participants who were exposed to study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 and 2 Pooled: NT 201 20 U | NT 201 50 U | NT 201 75 U | NT 201 100 U
Number analyzed (Participants) | 62 | 60 | 61 | 58
Participants | 25 | 23 | 26 | 22

3. Primary Outcome: Number of Participants With at Least One Treatment-emergent Serious Adverse Event (TESAE)
Time Frame: From the time of first treatment up to Day 390
Population: The SES was the subset of all participants who were exposed to study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 and 2 Pooled: NT 201 20 U | NT 201 50 U | NT 201 75 U | NT 201 100 U
Number analyzed (Participants) | 62 | 60 | 61 | 58
Participants | 0 | 0 | 0 | 1

4. Primary Outcome: Number of Participants With at Least One Treatment-emergent Adverse Event of Special Interest (TEAESI)
Time Frame: From the time of first treatment up to Day 390
Population: The SES was the subset of all participants who were exposed to study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 and 2 Pooled: NT 201 20 U | NT 201 50 U | NT 201 75 U | NT 201 100 U
Number analyzed (Participants) | 62 | 60 | 61 | 58
Participants | 1 | 0 | 2 | 2

5. Primary Outcome: Number of Participants With at Least One Treatment Related TEAE
Time Frame: From the time of first treatment up to Day 390
Population: The SES was the subset of all participants who were exposed to study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 and 2 Pooled: NT 201 20 U | NT 201 50 U | NT 201 75 U | NT 201 100 U
Number analyzed (Participants) | 62 | 60 | 61 | 58
Participants | 7 | 6 | 8 | 7

6. Primary Outcome: Number of Participants With at Least One Treatment Related TESAE
Time Frame: From the time of first treatment up to Day 390
Population: The SES was the subset of all participants who were exposed to study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 and 2 Pooled: NT 201 20 U | NT 201 50 U | NT 201 75 U | NT 201 100 U
Number analyzed (Participants) | 62 | 60 | 61 | 58
Participants | 0 | 0 | 0 | 0

7. Secondary Outcome: Duration of Effect Whereby Effect Was Defined as Score of None (0) or Mild (1) at Maximum Frown as Assessed by the Investigator According to FWS
Description: Duration of effect was defined as time between treatment and first point in time when score was moderate or severe again. If no effect was observed, duration of effect was set to 0. Effect was defined by a score of none (0) or mild (1) at maximum frown as assessed by investigator according to FWS. Investigator's FWS assessed status of GFL according to 4-point severity grades at maximum frown as: 0 (none), 1 (mild), 2 (moderate), 3 (severe). Descriptors of each severity grade for investigator's FWS assessment at maximum frown were as: 0 (no muscle action at all), 1 (some even slight muscle action possible [that is, visible furrows]), 2 (moderately strong muscle action possible [that is, visible muscle bulges]), 3 (strong muscle action possible which may cause local pallor). Duration of effect was analyzed using Kaplan-meier analysis, and 95% CI were calculated using log-log transformation.
Time Frame: From the time of first treatment up to Day 360
Population: The FAS was subset of participants exposed to study medication for whom any efficacy variable was available.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Stage 1 and 2 Pooled: NT 201 20 U | NT 201 50 U | NT 201 75 U | NT 201 100 U
Number analyzed (Participants) | 61 | 60 | 61 | 59
days | 113 [91 to 134] | 121 [113 to 149] | 129 [122 to 157] | 148 [125 to 173]

8. Secondary Outcome: Duration of Effect Whereby Effect Was Defined by 2-point Improvement From Baseline at Maximum Frown as Assessed by the Investigator According to FWS
Description: Duration of effect: time between treatment and first point in time when improvement was less than 2 points again. If no effect was observed, duration of effect was set to 0. Effect: at least a 2-point improvement from baseline at maximum frown as assessed by investigator on the FWS. Investigator's FWS assessed status of GFL according to 4-point severity grades at maximum frown as: 0 (none), 1 (mild), 2 (moderate), 3 (severe). Descriptors of each severity grade for investigator's FWS assessment at maximum frown were as: 0 (no muscle action at all), 1 (some even slight muscle action possible [that is, visible furrows]), 2 (moderately strong muscle action possible [that is, visible muscle bulges]), 3 (strong muscle action possible which may cause local pallor). Duration of effect was analyzed using Kaplan-meier analysis, and 95% CI were calculated using log-log transformation.
Time Frame: From the time of first treatment up to Day 360
Population: The FAS was subset of participants exposed to study medication for whom any efficacy variable was available.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Stage 1 and 2 Pooled: NT 201 20 U | NT 201 50 U | NT 201 75 U | NT 201 100 U
Number analyzed (Participants) | 61 | 60 | 61 | 59
days | 96 [90 to 118] | 118 [91 to 127] | 122 [119 to 127] | 145 [120 to 149]

9. Secondary Outcome: Percentage of Participants Rated as None (0) or Mild (1) at Maximum Frown by Investigator's Rating on FWS
Description: Investigator's FWS assessed status of GFL according to the 4-point severity grades at maximum frown as: 0 (none), 1 (mild), 2 (moderate), 3 (severe). Descriptors of each severity grade for investigator's FWS assessment at maximum frown were as: 0 (no muscle action at all), 1 (some even slight muscle action possible [that is, visible furrows]), 2 (moderately strong muscle action possible [that is, visible muscle bulges]), 3 (strong muscle action possible which may cause local pallor). 95% CIs for percentage of participants were based on Pearson-clopper method.
Time Frame: At Day 180
Population: The FAS was subset of participants exposed to study medication for whom any efficacy variable was available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1 and 2 Pooled: NT 201 20 U | NT 201 50 U | NT 201 75 U | NT 201 100 U
Number analyzed (Participants) | 61 | 60 | 61 | 59
percentage of participants | 8.2 [2.7 to 18.1] | 8.3 [2.8 to 18.4] | 16.4 [8.2 to 28.1] | 18.6 [9.7 to 30.9]

10. Secondary Outcome: Percentage of Participants Rated as None (0) or Mild (1) at Maximum Frown by Participant's Rating on FWS
Description: Participant's FWS assessed status of GFL according to the 4-point severity grades at maximum frown as: 0 (none), 1 (mild), 2 (moderate), 3 (severe). Descriptors of each severity grade for participant's FWS assessment at maximum frown were as: 0 (no muscle action at all), 1 (some even slight muscle action possible [that is, visible furrows]), 2 (moderately strong muscle action possible [that is, visible muscle bulges]), 3 (strong muscle action possible which may cause local pallor). 95% CI for percentage of participants were based on Pearson-clopper method.
Time Frame: At Day 180
Population: The FAS was subset of participants exposed to study medication for whom any efficacy variable was available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1 and 2 Pooled: NT 201 20 U | NT 201 50 U | NT 201 75 U | NT 201 100 U
Number analyzed (Participants) | 61 | 60 | 61 | 59
percentage of participants | 6.6 [1.8 to 15.9] | 10.0 [3.8 to 20.5] | 19.7 [10.6 to 31.8] | 16.9 [8.4 to 29.0]

11. Secondary Outcome: Percentage of Participants Rated as at Least 1-point Improvement Compared to Baseline at Maximum Frown by Investigator's Rating on FWS
Description: Investigator's FWS assessed status of GFL according to the 4-point severity grades at maximum frown as: 0 (none), 1 (mild), 2 (moderate), 3 (severe). Descriptors of each severity grade for investigator's FWS assessment at maximum frown were as: 0 (no muscle action at all), 1 (some even slight muscle action possible [that is, visible furrows]), 2 (moderately strong muscle action possible [that is, visible muscle bulges]), 3 (strong muscle action possible which may cause local pallor). 95% CI for percentage of participants were based on Pearson-clopper method.
Time Frame: At Day 180
Population: The FAS was subset of participants exposed to study medication for whom any efficacy variable was available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1 and 2 Pooled: NT 201 20 U | NT 201 50 U | NT 201 75 U | NT 201 100 U
Number analyzed (Participants) | 61 | 60 | 61 | 59
percentage of participants | 32.8 [21.3 to 46.0] | 43.3 [30.6 to 56.8] | 52.5 [39.3 to 65.4] | 52.5 [39.1 to 65.7]

12. Secondary Outcome: Percentage of Participants Rated as at Least 1-point Improvement Compared to Baseline at Maximum Frown by Participant's Rating on FWS
Description: as for outcome 10
Time Frame: At Day 180
Population: The FAS was subset of participants exposed to study medication for whom any efficacy variable was available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1 and 2 Pooled: NT 201 20 U | NT 201 50 U | NT 201 75 U | NT 201 100 U
Number analyzed (Participants) | 61 | 60 | 61 | 59
percentage of participants | 37.7 [25.6 to 51.0] | 36.7 [24.6 to 50.1] | 52.5 [39.3 to 65.4] | 45.8 [32.7 to 59.2]

ADVERSE EVENTS:
Time Frame: From the time of first treatment up to Day 390
Description: As planned, combined safety data for NT 201 administered in MP and OLEX were reported.
Arm/Group | Stage 1 and 2 Pooled: NT 201 20 U | NT 201 50 U | NT 201 75 U | NT 201 100 U
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/60 | 0/61 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/60 | 0/61 | 1/58
Other Adverse Events (participants affected / at risk) | 13/62 | 11/60 | 12/61 | 12/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1 and 2 Pooled: NT 201 20 U (N=62) | NT 201 50 U (N=60) | NT 201 75 U (N=61) | NT 201 100 U (N=58)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1 and 2 Pooled: NT 201 20 U (N=62) | NT 201 50 U (N=60) | NT 201 75 U (N=61) | NT 201 100 U (N=58)
Headache (Nervous system disorders) | 6 (8) | 6 (8) | 1 (1) | 4 (4)
Nasopharyngitis (Infections and infestations) | 11 (14) | 6 (7) | 11 (11) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.

DOCUMENTS (2):
  • Study Protocol (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT03806933/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/33/NCT03806933/SAP_001.pdf